CLINICAL TRIAL: NCT04172883
Title: Management of Device Detected Atrial Tachyarrhythmia( AT) and Impact of Device Treatment Algorithms on Atrial Fibrillation (AF) in Indian Population
Brief Title: Management of Device Detected AT and Impact of Device Treatment Algorithms on Atrial Fibrillation
Acronym: MANDATE-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MDT18039
Record Dates: First submitted 2019-05-28; First posted 2019-11-21 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Cardiovascular Diseases
Keywords: Reactive ATP; device based Management of Atrial fibrilation; AF Management
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient is unaware of which type of programming changes have been made ( whether it is the reduced sequence programming or the standard Minerva setting )
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): The devices on the study are all commercially available and enabled with reactive ATP( rATP)feature, for the study both arms will have rATP switched on with one arm on the standard device setting or MINERVA setting ( control arm)
- Treatment arm (Active Comparator): The devices on the study are all commercially available and enabled with reactive ATP( rATP)feature, for the study both arms will have rATP switched on with one arm on the reduced sequence programming ( treatment arm)
  Interventions: Other: Treatment arm

INTERVENTIONS:
Other: Treatment arm — All pts are implanted with rATP enabled devices prior to the study start , the only intervention in both arms is switching on rATP and in the treatment arm programming changes done to optimize the rATP sequence delivery of therapy and prevent the patient from going into permanent or persistent AF
  Other Names: programming changes
  Arms: Treatment arm

SUMMARY:
The MANDATE-AF study was designed to address evidence needs in India for device-based management of AF using AT/AF (Atrial Tachycardia/Atrial fibrillation) diagnostic features and therapies such as Reactive Atrial anti tachycardia Pacing (rATP) within Medtronic Cardiac Implantable Electronic Devices (CIED)and its impact on the time to persistent AF and progression of AT/AF.

DETAILED DESCRIPTION:
New generation Cardiac Implantable Electronic devices (CIED's)such as Pacemakers, Implantable Cardioverter Defibrillator (ICD) and Cardiac Resynchronization Therapy (CRT) has diagnostic and treatment delivery features which helps in slowing the progression of Atrial Fibrillation. A Study conducted in Europe, called the MINERVA Trial, showed the efficacy of a feature within Medtronic CIED's called (rATP)™, in the termination of abnormal rhythms by pacing stimuli, and clinical benefit in reducing incidence of Atrial Fibrillation. However, there is dearth of local evidence of this within the Indian population and also a need to show that turning on rATP does not compromise on battery depletion.

The MANDATE-AF study is a prospective , Interventional , Randomized, single blind study aiming to show that a reduced sequence programming of this rATP therapy ,can improve device battery longevity and is as effective as the Minerva trial ATP programming when it comes to showing its impact on time to persistent AF and on the progression of AT/AF within the Indian population.

The study analyses patients implanted with a Medtronic cardiac implantable device with an atrial lead and equipped with atrial ATP therapies.

The patients will be randomized into two groups:

* an interventional arm including patients with a conservative atrial ATP therapies programming setting
* a control, arm including patients with the same atrial ATP therapies programming setting adopted in the Minerva Trial

Cardiovascular events will be collected prospectively for at least 24 months after enrollment. Physicians will be recommended to schedule in clinic follow-up visits every 6 months and remote follow-up visits every 3 months in between. Every patient will be followed for at least 24 months, until the last patient enrolled exits the study.

ELIGIBILITY:
Inclusion Criteria:

1 Subject is implanted with a Medtronic cardiac implantable device with an atrial lead equipped with atrial ATP therapies (rATP) enabled no longer than 18 months and at the minimum 6 weeks has passed since the implant; 2. Age > 55 years; 3. Subject provides informed consent; 4. Subject is willing and able to comply with the study procedures; 5. Subject has documented history of atrial fibrillation or atrial flutter, or one or more of the risk factors for developing AF as per AHA/HRS (American heart Association/Heart rhythm Society) guidelines.

* Age > 60 years;
* Stroke/TIA (Transient ischemic Attack);
* Diabetes;
* High Blood Pressure;
* Coronary artery disease;
* Cardiomyopathy;
* Pericardial inflammation;
* Prior heart attacks;
* Congestive heart failure;
* Structural heart disease (valve problems or congenital defects);
* Prior open-heart surgery;
* Untreated atrial flutter (another type of abnormal heart rhythm);
* Thyroid disease;
* Chronic lung disease;
* Sleep apnea;
* Excessive alcohol use;
* Serious illness or infection.

Exclusion criteria:

Patients are not eligible to be enrolled in the study if any of the following criteria is met:

1. Subject has been implanted with a Medtronic cardiac implantable device with an atrial lead equipped with atrial ATP therapies (rATP) enabled for more than 18 months;
2. Subject is in permanent AF or persistent AF at the baseline visit:

   1. The definition of permanent AF will be based on the physicians' decision that nothing further can be done to cardiovert the patient or, in historical cases, the investigators will refer to the Cardiac Compass reports:
   2. The definition of persistent AF at baseline will refer to the Cardiac Compass reports (>7 consecutive days in AF with the last day being the day of enrollment)
3. Participation in other studies which could potentially conflict with this study;
4. Legal incapacity or evidence that a subject cannot understand the purpose and risks of the study or inability to comply fully with study procedures and follow up.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Time to persistent AF | 42months
  time to persistent AF (defined as more than 7 continuous days of AF) or permanent AF

SECONDARY OUTCOMES:
All-cause death(at the end of 24 months) | 42months
  Compare the two atrial ATP Programming arms in terms of clinical endpoints such as deaths that occur on the study
Number of Cardiovascular hospitalization | 42 Months
  Compare the two atrial ATP Programming arms in terms of clinical endpoints such as cardiovascular hospitalizations (due to Heart Failure (HF), AF or other), as measured by the time to first event and annual rate of such events
Annual rate for all-cause hospitalization | 42 months
  Compare the two atrial ATP Programming arms in terms of clinical endpoints such as all cause hospitalizations and its annual rate on the study
Measure the AT/AF burden metrics across various time points | 42 months
  Compare the two atrial ATP Programming arms in terms of clinical endpoints to evaluate the AT/AF burden metrics (amount of time each AF event lasts) as measured in terms of time to first event (daily burden ≥1 day, ≥2 days, ≥30 days) or the ratio between time in AT/AF and the observation period (the duration the patient is on the study)
Evaluate number of successful and unsuccessful treated AT/AF episodes out of the detected episodes | 42 months
  Compare the two atrial ATP Programming arms in terms of clinical endpoints to assess number of successful and unsuccessful treated AT/AF episodes out of detected episodes by the device .
Measure number of delivered therapies per episode | 42 months
  compare the two atrial ATP Programming arms in terms of clinical endpoints to measure the number of therapies delivered per episode to mitigate the AT/AF event.
Evaluate the number of ATP sequences | 42 months
  Compare the two ATP programming arms in terms of clinical endpoints to measure the number of ATP sequences delivered on each arm.
Evaluate number of stroke, TIA (Transient ischemic Attack ) or other thromboembolic events | 42 months
  compare the two atrial ATP Programming arms in terms of clinical endpoints to calculate number of stroke, TIA or other thromboembolic events reported on the study across both arms
Percentage of patients treated with anticoagulation therapy | 42 months
  Compare the two ATP programming arms in terms of clinical endpoints to evaluate the percentage of patients treated with anticoagulation therapy according to AF management guideline
Measure the LA diameter size | 42 months
  Compare the two ATP programming arms in terms of clinical endpoints to evaluate the LA diameter (if available) as measured through an Echocardiogram
Number of Pharmacological and electrical cardio versions reported | 42 months
  Compare the two ATP programming arms in terms of clinical endpoints such as number of electrical or pharmacological cardio-versions measured in terms of time to first event and its annual rate on the study;
Evaluate the biventricular pacing percentage | 42 months
  Compare the two ATP programming arms in terms of clinical endpoints such as biventricular pacing percentage (in cardiac resynchronization therapy defibrillator (CRT-D) / cardiac resynchronization therapy-Pacemaker (CRT-P) patients)
Incidence of the composite endpoints like death or Cardiovascular Hospitalizations | 42months
  A cumulative endpoint which includes number of deaths, cardiovascular hospitalizations, stroke, TIA or other thromboembolic events.
Incidence of persistent AF in patients with sick sinus syndrome | 42 months
  To evaluate the incidence of persistent AF in patients with sick sinus syndrome as compared to the one found in the Minerva trial, and characterize the difference between the European and Indian populations. The unit of measure will be number of pts that had persistent AF on the study.
Efficacy of Atrial ATP therapies measured by number of successful termination of AF events | 42 months
  To evaluate the efficacy of atrial ATP therapies as a function of the device type (Pacemakers(IPG),Cardiac defibrillators (ICD),Cardiac resynchronization Therapy (CRT-D, CRT-P), and population characteristics (baseline characteristics, implant indications) in optimizing therapy and evaluating the successful termination of AF events, preventing pts from going into persistent or permanent AF, as measured by no of ATP's delivered by device.

CONTACTS AND LOCATIONS:
Overall Officials: Shantanu Sarkar, PhD, Study Chair — Medtronic, PLC
Locations (11):
- India (11):
  - Care Institute of medical sciences and research, Ahmedabad, Gujarat
  - Apollo Hospital , Bannerghatta, Bangalore, Karnataka
  - Apollo BGS Hospital, Mysore, Karnataka
  - Aster Medicity, Kochi, Kerala
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Fortis Escorts Heart Institute, New Delhi, National Capital Territory of Delhi
  - Apollo Hospital, Bhubaneshwar, Odisha
  - Fortis Escort Hospital, Mohali, Punjab
  - Eternal Heart Care center and Research, Jaipur, Rajasthan
  - Apollo Hospital, Chennai, Tamil Nadu
  - AIG hospital, Hyderabad, Telangana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stewart S, Hart CL, Hole DJ, McMurray JJ. A population-based study of the long-term risks associated with atrial fibrillation: 20-year follow-up of the Renfrew/Paisley study. Am J Med. 2002 Oct 1;113(5):359-64. doi: 10.1016/s0002-9343(02)01236-6. PMID 12401529
- [Result] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Result] Camm AJ, Kirchhof P, Lip GY, Schotten U, Savelieva I, Ernst S, Van Gelder IC, Al-Attar N, Hindricks G, Prendergast B, Heidbuchel H, Alfieri O, Angelini A, Atar D, Colonna P, De Caterina R, De Sutter J, Goette A, Gorenek B, Heldal M, Hohloser SH, Kolh P, Le Heuzey JY, Ponikowski P, Rutten FH; ESC Committee for Practice Guidelines. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). Europace. 2010 Oct;12(10):1360-420. doi: 10.1093/europace/euq350. No abstract available. PMID 20876603
- [Result] Kannel WB, Wolf PA, Benjamin EJ, Levy D. Prevalence, incidence, prognosis, and predisposing conditions for atrial fibrillation: population-based estimates. Am J Cardiol. 1998 Oct 16;82(8A):2N-9N. doi: 10.1016/s0002-9149(98)00583-9. PMID 9809895